CLINICAL TRIAL: NCT01207297
Title: Tacrolimus Versus Cyclophosphamide as Treatment for Diffuse Proliferative or Membranous Lupus Nephritis: Prospective Cohort Study
Brief Title: Tacrolimus Versus Cyclophosphamide as Treatment for Lupus Nephritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Jianghua Chen, Tacrolimus versus cyclophosphamide as treatment for diffuse proliferative or membranous lupus nephritis: prospective cohort study, Zhejiang University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChiCTR-TKMS-1000960; ChiCTR-TNRC-10000960 (Other: Chinese Clinical Traial Registry)
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2010-09

CONDITIONS: SLE; Lupus Nephritis; Renal Insufficiency; End-stage Renal Disease
Keywords: Lupus nephritis; tacrolimus; cyclophosphamide
MeSH Terms: conditions — Lupus Nephritis; Renal Insufficiency; Kidney Failure, Chronic | interventions — Tacrolimus; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAC group (Active Comparator): Oral tacrolimus (0.04-0.08 mg/kg/d) and prednisone for 12 months.
  Interventions: Drug: Tacrolimus
- CYC group (Active Comparator): Pulse cyclophosphamide (750mg/m2 per month for six months) and prednisone followed by azathioprine (50mg/day）for 6 months.
  Interventions: Drug: cyclophosphamide

INTERVENTIONS:
Drug: Tacrolimus — The calcineurin inhibitor is widely administered for organ transplantation，which establish the current method for lupus nephritis (LN).
  20 patients with LN were self-assigned the therapy of TAC and prednisone for 12 months. The dosage was adjusted to achieve a whole blood TAC 12 h trough concentration.
  Other Names: Prograf
  Arms: TAC group
Drug: cyclophosphamide — 20 patients with LN were self-assigned the protolcol of intravenous cyclophosphamide (750mg/m2 per month)/prednisone for six months followed by azathioprine(100mg/day)/prednisone for six months.
  Arms: CYC group

SUMMARY:
In this comparative open-label cohort study, the investigators compared the efficacy and safety of tacrolimus (TAC)and cyclophosphamide (CYC) in the treatment of diffuse proliferative and membranous lupus nephritis with severe renal disease. Treatment of lupus nephritis (LN) with cyclophosphamide is effective, but retain a certain proportion of renal function exacerbations. Tacrolimus may be a suitable substitute treatment for CYC.

Methods: Forty patients with diffuse proliferative or membranous were recruited for this trial, 45% of them had lower Ccr (<60mL/min/1.73m2), 10% had increased serum creatinine (>180µmol/L) and 67.5% had nephritic proteinuria (>3.5g/day). The investigators compared the efficacy and adverse effects of TAC (0.04-0.08 mg/kg/d) and prednisone for 12 months (TAC group) with pulse cyclophosphamide (750mg/m2 per month for six months) and prednisone followed by azathioprine (50mg/day）for 6 months (CYC group).

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a multisystem autoimmune disease. About 60% of SLE patients have renal disease, and patients with rapidly progressive destruction of renal parenchyma have significantly poorer prognosis. Drug therapies that employ corticosteroids, cyclophosphamide, and/or mycophenolate mofetil have improved patient outcomes, but a significant number of patients have refractory disease or cannot tolerate these drugs. Moreover, SLE patients who are partially responsive or resistant to treatment have significant morbidity，mortality, and exacerbations of renal function. Thus, in patients with lupus nephritis (LN), the two main causes of morbidity and mortality are treatment-related or patient-related. It has been suggested that new therapies be developed for SLE that more specifically target the relevant immunopathogenetic pathways, so as to achieve greater efficacy and reduce therapy-related toxicities ，and to save or protect renal function.

Tacrolimus (TAC) is an immunosuppressive macrolide of the calcineurin inhibitor (CNI) group that is widely administered following organ transplantation. In 1989, Takabayashi K. et al. studied the effect of TAC on a murine model of SLE, and showed that it prolonged lifespan, reduced proteinuria, and prevented the progression of nephropathy, although it had no appreciable effect on the levels of anti-dsDNA antibodies. More recent small-scale studies have shown that TAC may be an effective treatment for nephritic syndrome and LN8-11. However, there is little clinical experience in the use of TAC for treatment of LN, especially for LN with severe renal disease, and limited knowledge of the comparative efficacy of TAC and other therapies.

In this comparative open-label cohort study, we compared the efficacy and safety of TAC and CYC in the treatment of diffuse proliferative and membranous lupus nephritis with severe renal disease.

LN is characterized by autoantibody-mediated vasculitis that may lead to rapid progression of multi-system and organ damage. The kidneys are often involved due to excretion of excessive urinary protein and/or rapidly progressive kidney injury, and end-stage renal disease may result. Treatment-related differences in the rates of renal failure may not be discernible early in the course of treatment, but there are definite advantages of rapid remission, effective prophylaxis against relapse, and prevention of renal failure.

An intravenous pulse CYC regime has been the "gold standard" immunosuppressive regime for the treatment of LN. The activation of lymphocytes, production of autoantibody, and high expression of IFN-γ in the circulation and renal tissue are important indicators of renal injury in SLE. Previous clinical and animal studies have shown that TAC therapy inhibits T-lymphocyte activation, suppresses cytokine production in lymphocytes, suppresses antigen-induced monokine (TNF-α) production in macrophages, reduces interleukin-2 mRNA expression, decreases serum levels of IFN-γ and IFN-γ mRNA expression in the kidney and spleen, and decreases serum levels of IgG-class anti-DNA antibodies. A recent study also showed that TAC treatment affects B-cell antibody responses indirectly by interfering with T-helper cells.

The risk of end-stage renal failure is particularly high in patients with diffuse proliferative glomerulonephritis. Despite the diverse and complex interplay of various causative factors in individual patients, two previous studies suggested that SLE patients who experience glomerulonephritis that does not diminish following treatment with conventional immunosuppressive therapies have increased risk for subsequent deterioration of renal function and poor long-term outcome. This suggests that there is an urgent need for alternative immunosuppressive therapies for treatment of SLE, and motivated our investigation of TAC. On the other hand, it is well know that calcineurin inhibitors (such as TAC) are associated with chronic nephrotoxicity. For example, Tse et al. showed that one of six patients developed chronic nephrotoxicity after 10 months of TAC therapy. As a calcineurin inhibitor, TAC has a lower potential for nephrotoxicity than cyclosporine.

Opportunistic infection is a severe complication that can result from treatment of LN with immunosuppressive drugs.

ELIGIBILITY:
Inclusion Criteria:

* SLE patients:diagnosis based on American Rheumatism Association criteria;
* renal biopsy-proven active LN (diffuse proliferative and membranous lupus nephritis, class IV, V, V+IV and/or V+III, according to the ISN/RPS 2003 classification13)
* urinary protein excretion of at least 2.0 g per 24 h
* serum creatinine less than 221 µmol/dL (2.5mg/dL)
* creatinine clearance more than 30 mL/min/1.73m2

Exclusion Criteria:

* pregnant or lactating
* previous treatment with cyclosporine, mycophenolate mofetil treatment for at least two weeks in the previous three months
* known allergies to calcineurin inhibitors
* severe infection or illness
* symptoms of a central nervous system disorder
* alanine aminotransferase more than 100U/L
* evidence of active hepatitis
* fasting blood glucose more than 6.2 mmol/L
* 2 h post-meal blood glucose more than 11.1mmol/L

Ages: 15 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2003-03; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Tacrolimus versus cyclophosphamide as treatment for diffuse proliferative or membranous lupus nephritis | one year
  The primary study outcome measure was the cumulative rate of complete remission (CR).

SECONDARY OUTCOMES:
Evaluating the effective and safety of TAC for severe lupus nephritis compared CYC protocol. | one year
  The secondary outcome measure were time required for CR, cumulative rate of sustained remission, relapse rate, immunological parameters, side effects, renal function during treatment and followed-up, and compliance with therapy and TAC dosing and serum levels.

CONTACTS AND LOCATIONS:
Overall Officials: Jianghua Chen, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University